CLINICAL TRIAL: NCT06209203
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase II Clinical Trial to Evaluate the Efficacy and Safety of ZKY001 Eye Drops in Patients with Corneal Epithelial Defects After TPRK
Brief Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of ZKY001 Eye Drops
Acronym: TPRK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKO-SFT-202112-TPRK
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-01

CONDITIONS: Corneal Epithelium Defect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lowe-dose ZKY001 eye drops (Experimental): The drug was given once immediately after surgery on D0, and 1 drop was given 4 times a day from D0 to D6
  Interventions: Drug: lowe-dose ZKY001 eye drops
- Medium-dose ZKY001 eye drops (Experimental): The drug was given once immediately after surgery on D0, and 1 drop was given 4 times a day from D0 to D6
  Interventions: Drug: Medium-dose ZKY001 eye drops
- placebo (Placebo Comparator): The drug was given once immediately after surgery on D0, and 1 drop was given 4 times a day from D0 to D6
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lowe-dose ZKY001 eye drops — eye drops
  Other Names: ZKY001
  Arms: lowe-dose ZKY001 eye drops
Drug: Medium-dose ZKY001 eye drops — eye drops
  Other Names: ZKY001
  Arms: Medium-dose ZKY001 eye drops
Drug: placebo — eye drops
  Other Names: Simulated eye drops
  Arms: placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled clinical trial was designed. A total of 120 subjects were randomly assigned to two experimental groups (lowe-dose ZKY001 eye drops group,Medium-dose ZKY001 eye drops group) and a placebo control group, with 40 subjects in each group.

DETAILED DESCRIPTION:
Study cycle: 7 days screening period (d-7-D-1), 7 days treatment period (D0-D6), and the end of the study on D7.

Statistical analysis was performed using SAS9.4 or above software. All statistical tests were two-sided, and P less than or equal to 0.05 was considered statistically significant for the difference being tested unless specified.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-40 years old, regardless of gender;
2. Plan TPRK for myopia and/or myopic astigmatism, meet the indications for TPRK, and set the ablation diameter of the optical zone at 6.0-6.5 mm;
3. Schirmer test I ≥10mm/5min;

Exclusion Criteria:

1. prior corneal refractive surgery or keratoplasty;
2. Contraindications to TPRK surgery, including severe ocular surface disease that may affect the corneal epithelium, active ocular inflammation, moderate to severe dry eye, keratoconus or other types of corneal ectasia, thin corneas, severe lesions of ocular appendages (such as eyelid defects, deformations, etc.), glaucoma, cataract that affects vision, History of systemic immune diseases (systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, etc.);
3. incomplete eyelid closure;
4. corneal degeneration, corneal stroma or endothelial damage or malnutrition;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
healing time | seven days
  Corneal epithelial healing time

SECONDARY OUTCOMES:
number of healing | seven days
  The percentage of corneal healing at 24h, 48h, 72h, 120h and 168h after operation

OTHER OUTCOMES:
Corneal staining | seven days
  The percentage of corneal staining negative at 48h, 72h, 120h and 168h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xingtao Zhou, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China